CLINICAL TRIAL: NCT00851721
Title: FEIBA NF: A Prospective, Open-label, Randomized, Parallel Study to Evaluate the Efficacy and Safety of Prophylactic Versus On-Demand Treatment in Subjects With Hemophilia A or B and a High Titer Inhibitor
Brief Title: Efficacy and Safety Study of Prophylactic Versus On-Demand Treatment With Feiba NF in Subjects With Hemophilia A or B and a High Titer Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090701; 2008-003855-65 (EudraCT Number)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A or B With Inhibitors; Hemophilia A; Hemophilia B
Keywords: Hemophilia A; Factor VIII Inhibitor; Factor IX Inhibitor; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis arm (Experimental)
  Interventions: Biological: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated)
- On-demand arm (Active Comparator)
  Interventions: Biological: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated)

INTERVENTIONS:
Biological: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) — 85 ± 15 U/kg of FEIBA NF every other day during the 12-month prophylactic period
  Other Names: FEIBA NF
  Arms: Prophylaxis arm
Biological: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) — FEIBA NF dose and dosing interval as prescribed by the treating physician
  Other Names: FEIBA NF
  Arms: On-demand arm

SUMMARY:
The purpose of the study was to determine the efficacy, safety, and health-related quality of life benefits with FEIBA NF prophylactic treatment as compared with on-demand treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form by the participant or the participant's legally authorized representative
* The participant is ≥ 4 to ≤ 65 years of age
* The participant has a Karnofsky performance score of ≥ 60
* Hemophilia A and B of any severity, with documented history of high-titer inhibitor (> 5 Bethesda unit (BU)) for at least 12 months; or, if inhibitor titer is ≤ 5 BU, and the participant is refractory with increased dosing of either factor VIII (FVIII) or factor IX (FIX), as demonstrated from the participant's medical history
* Currently being treated on an on-demand basis for treatment of bleeding episodes
* Adequate venous access, with or without central venous device
* ≥ 12 bleeding episodes requiring treatment with by-passing agents in the past 12 months, based on medical history
* Competent in-home treatment and infusion therapy
* Currently using bypassing agents (activated prothrombin complex concentrate (APCC) or recombinant activated factor VII (rFVIIa)) for treatment of bleeding episodes
* HCV-, either by antibody testing or polymerase chain reaction (PCR); or HCV+ with stable hepatic disease
* HIV-, or HIV+ with stable disease and CD4 count > 200 cells/mm3 at screening
* Female participant of childbearing potential, presents with a negative serum pregnancy test, and agrees to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Currently receiving immune tolerance induction (ITI)
* Currently on regular prophylactic therapy to prevent bleeding episodes
* Clinically symptomatic liver disease (e.g. diagnosis of cirrhosis [confirmed by liver biopsy], portal vein hypertension, ascites, prothrombin time (PT) 5 seconds above upper limit of normal)
* Platelet count < 100,000/ml
* Planned elective surgery during participation in this study
* Participant is currently participating in another clinical study and has received an investigational product or device within 30 days prior to study entry
* Planned use of pegylated or non-pegylated alpha-interferon with or without ribavirin for HCV infected participants or planned use of a protease inhibitor for HIV infected participants. Participants currently taking any of these medications for a 30-day course are eligible.
* Clinically significant increase in D-dimer levels from historical baseline and/or associated with chronic liver disease or clinically evident thromboembolic event
* Known hypersensitivity to anti-inhibitor coagulant complexes (AICCs)
* Currently treated with a systemic immunomodulating drug
* Prior history of thromboembolic event: acute myocardial infarction, deep vein thrombosis, or pulmonary embolism
* Diagnosis of advanced atherosclerosis, malignancy and/or other diseases that may increase the participant's risk of thromboembolic complications
* Clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03-31 (Actual); Primary Completion 2012-10-17 (Actual); Study Completion 2012-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (2):
  - Chicago, Illinois
  - Cleveland, Ohio
- Brazil (2):
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
- Sofia, Bulgaria
- Zagreb, Croatia
- Japan (2):
  - Kanagawa
  - Nara
- Wellington, New Zealand
- Poland (2):
  - Krakow
  - Warsaw
- Romania (2):
  - Bucharest
  - Timișoara
- Russia (3):
  - Kirov
  - Moscow
  - Yekaterinburg
- Lviv, Ukraine

REFERENCES:
- [Result] Antunes SV, Tangada S, Stasyshyn O, Mamonov V, Phillips J, Guzman-Becerra N, Grigorian A, Ewenstein B, Wong WY. Randomized comparison of prophylaxis and on-demand regimens with FEIBA NF in the treatment of haemophilia A and B with inhibitors. Haemophilia. 2014 Jan;20(1):65-72. doi: 10.1111/hae.12246. Epub 2013 Aug 1. PMID 23910578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted in Europe, North America, Asia-Pacific, and South America at 17 clinical sites beginning in March 2009.
Pre-assignment Details: 52 participants were enrolled. Sixteen participants discontinued, (ten were screen failures and six were withdrawn before randomization (2 sponsor's decision- inhibitors, 3 withdrew consent, and 1 due to investigator decision to have participant on prophylaxis). Therefore 36 participants were randomized.
Groups:
- On-demand Arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : Standard FEIBA NF dose and dosing interval as prescribed by the treating physician
- Prophylaxis Arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : 85 ± 15 U/kg of FEIBA NF every other day during the 12-month prophylactic period
Period: Overall Study
Arm/Group | On-demand Arm | Prophylaxis Arm
Started | 19 | 17
Completed | 17 | 16
Not Completed | 2 | 1
Not completed — planned surgery | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-demand Arm | Prophylaxis Arm | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (15.2) | 25.6 (15.4) | 27.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 17 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
  Poland | 1 | 1 | 2
  Brazil | 3 | 2 | 5
  Ukraine | 4 | 4 | 8
  Romania | 0 | 1 | 1
  Croatia | 0 | 1 | 1
  Russian Federation | 8 | 3 | 11
  Bulgaria | 0 | 2 | 2
  Japan | 1 | 1 | 2
  New Zealand | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Annualized Bleeding Episode Rate (ABR) Among Participants Receiving Prophylactic Treatment as Compared to Those Treated On-demand
Description: Participants were Randomized to Receive 1 of the 2 Following Treatment Regimens: 1.On-Demand: FEIBA NF dose & dosing interval as prescribed by treating physician 2.Prophylaxis: 85 ± 15 U/kg of FEIBA NF every other day during 12-month prophylactic period Annualized rate of bleeding episodes was calculated as: (Number of bleeding episodes/observed treatment period in days) * 365.25
Time Frame: 12 months ± 14 days
Population: Efficacy Intent to Treat Analysis Dataset: Dataset consists of data from all randomized participants. Dataset includes those who discontinued FEIBA NF but did not withdraw informed consent and were willing to continue providing data. For these participants, only the data collected before FEIBA NF discontinuation is included.
Measure: Median (Inter-Quartile Range); unit: bleeds/year
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
bleeds/year | 28.7 (1.8) [17.7 to 50.0] | 7.9 (1.8) [2.9 to 11.0]
Statistical Analysis 1: Comparison: On-demand Arm vs Prophylaxis Arm; H0: μ(on-demand) = μ(prophylaxis) Versus H1: μ(on-demand) ≠ μ(prophylaxis) (Where H0 implies no difference in mean bleeding episode rate between prophylaxis and on-demand treatment arms and H1 implies otherwise. This test was performed at a significance level of 5%, two-sided, two sample); Test type: Superiority or Other; p = 0.0003, Two-sample, two-sided t-test

2. Secondary Outcome: Annualized Bleeding Rate by Treatment Regimen, Bleeding Etiology, and Bleed Type
Description: Spontaneous includes unknown/undermined etiology
Time Frame: 12 months ± 14 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
Bleeds per year
  Spontaneous | 18.9 [10.9 to 43.5] | 5.6 [2.9 to 8.0]
  Traumatic | 4.7 [1.9 to 10.7] | 2.5 [0.0 to 3.1]
  Joint | 22.9 [14.1 to 46.9] | 6.0 [2.9 to 10.0]
  Non-Joint | 2.9 [1.0 to 4.9] | 0.5 [0.0 to 2.0]
  Spontaneous Joint | 16.6 [9.9 to 40.8] | 4.5 [2.9 to 8.0]
  Spontaneous Non-Joint | 1.0 [1.0 to 2.9] | 0.0 [0.0 to 1.0]
  Traumatic Joint | 4.0 [1.0 to 7.1] | 1.0 [0.0 to 3.1]
  Traumatic Non-Joint | 0.0 [0.0 to 1.9] | 0.0 [0.0 to 1.0]
  All Bleeding Etiologies, and Bleed Types | 28.7 [17.7 to 50.0] | 7.9 [2.9 to 11.0]

3. Secondary Outcome: Differences in Mean Transformed Annualized Bleeding Rate Between On-Demand and Prophylaxis Treatment Regimens by Bleeding Etiology, and Bleeding Type
Description: Annualized bleed rates were transformed using the square root of the number of bleeding episodes observed (X bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using the t-test. The difference in mean transformed ABRs was used to perform statistical tests and generate p-values at a significance level of 5% Participants were Randomized to Receive 1 of the 2 Following Treatment Regimens: 1.On-Demand: FEIBA NF dose & dosing interval as prescribed by treating physician 2.Prophylaxis: 85 ± 15 U/kg of FEIBA NF every other day during 12-month prophylactic period
Time Frame: 12 months ± 14 days
Population: Efficacy Intent to Treat Analysis Dataset
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- On-demand Arm Versus Prophylaxis Arm: On-demand arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : FEIBA NF dose and dosing interval as prescribed by the treating physician Prophylaxis arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : 85 ± 15 U/kg of FEIBA NF every other day during the 12-month prophylactic period
Arm/Group | On-demand Arm Versus Prophylaxis Arm
Number analyzed (Participants) | 36
(bleeds/year)^(1/2)
  Spontaneous Bleeds | 2.2 (1.8)
  Traumatic Bleeds | 1.0 (1.2)
  Joint Bleeds | 2.4 (1.9)
  Non-Joint Bleeds | 0.8 (0.9)
  Spontaneous Joint Bleeds | 2.1 (1.8)
  Spontaneous Non-Joint Bleeds | 0.8 (0.8)
  Traumatic Joint Bleeds | 0.9 (1.2)
  Traumatic Non-Joint Bleeds | -0.0 (0.9)
Statistical Analysis 1: Comparison: On-demand Arm Versus Prophylaxis Arm; Spontaneous Bleeds; Test type: Superiority or Other; p = 0.0008, Two-sample, two-sided t-test
Statistical Analysis 2: Comparison: On-demand Arm Versus Prophylaxis Arm; Traumatic Bleeds; Test type: Superiority or Other; p = 0.0199, Two-sample, two-sided t-test
Statistical Analysis 3: Comparison: On-demand Arm Versus Prophylaxis Arm; Joint Bleeds; Test type: Superiority or Other; p = 0.0006, Two-sample, two-sided t-test
Statistical Analysis 4: Comparison: On-demand Arm Versus Prophylaxis Arm; Non-Joint Bleeds; Test type: Superiority or Other; p = 0.0227, Two-sample, two-sided t-test
Statistical Analysis 5: Comparison: On-demand Arm Versus Prophylaxis Arm; Spontaneous Joint Bleeds; Test type: Superiority or Other; p = 0.0013, Two-sample, two-sided t-test
Statistical Analysis 6: Comparison: On-demand Arm Versus Prophylaxis Arm; Spontaneous Non-Joint Bleeds; Test type: Superiority or Other; p = 0.0030, Two-sample, two-sided t-test
Statistical Analysis 7: Comparison: On-demand Arm Versus Prophylaxis Arm; Traumatic Joint Bleeds; Test type: Superiority or Other; p = 0.0254, Two-sample, two-sided t-test
Statistical Analysis 8: Comparison: On-demand Arm Versus Prophylaxis Arm; Traumatic Non-Joint Bleeds; Test type: Superiority or Other; p = 0.9322, Two-sample, two-sided t-test

4. Secondary Outcome: Annualized Bleeding Rate for New Target Joints
Description: Target joints are ≥4 bleeds/6 months in any one of the following joints: ankles, knees, elbows, and hips; a target joint bleeding episode refers to an individual anatomical location.
Time Frame: 12 months ± 14 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
Bleeds per year | 5.9 [0.0 to 12.9] | 0.0 [0.0 to 4.1]

5. Secondary Outcome: Differences in Mean Transformed Annualized Bleeding Rate Between On-Demand and Prophylaxis Treatment Regimens: New Target Joints
Description: Annualized bleed rates (ABRs) were transformed using the square root of the number of bleeding episodes observed (X bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using a two-sample, two-sided t-test. The difference in mean transformed ABRs was used to perform statistical tests and generate p-values at a significance level of 5%
Time Frame: 12 months ± 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- On-demand Arm Versus Prophylaxis Arm: On-demand arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated): FEIBA NF dose and dosing interval as prescribed by the treating physician Prophylaxis arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : 85 ± 15 U/kg of FEIBA NF every other day during the 12-month prophylactic period
Arm/Group | On-demand Arm Versus Prophylaxis Arm
Number analyzed (Participants) | 36
(bleeds/year)^(1/2) | 1.6 (2.2)
Statistical Analysis 1: Comparison: On-demand Arm Versus Prophylaxis Arm; Test type: Superiority or Other; p = 0.0271, Two-sample, two-sided t-test

6. Secondary Outcome: Number of New Target Joints
Description: Target Joints are defined as ≥4 bleeds/6 months in any one of the following joints: ankles, knees, elbows and hips
Time Frame: 12 months ± 14 days
Population: as for outcome 1
Measure: Number; unit: new target joints
Groups:
- On-demand Arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : FEIBA NF dose and dosing interval as prescribed by the treating physician
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
new target joints | 23 | 7

7. Secondary Outcome: Assessment of Objective Clinical Symptoms- Visual Analog Scale (VAS): Pain in Adolescents and Adults (≥12 Years Old)
Description: Pain caused by a bleeding episode in adolescents and adults (≥12 years old) was measured at pre-infusion (pre-inf) and at 6 ± 0.5 hours (h) and 24 ± 1 h post-infusion (post-inf) (after the last infusion given to treat a bleeding episode) on the VAS pain scale in millimeters from 0 (no pain) to 100 (worst possible pain). For analysis purposes, if short acting analgesics (duration of activity approximately 6 ± 0.5 h) were used, pain was assigned the highest possible score (100). Pain assessment occurred after each infusion related to single bleeding episodes. In case participants required an additional infusion within 24h, pain was assessed 6 ± 0.5 h and 24 ±1 h following the subsequent infusion. Change in VAS scores at 6 ± 0.5 h and 24 ±1 h post-infusion were also compared relative to pre-infusion VAS scores (ie, (pre-infusion VAS score) - (post-infusion VAS score)).
Time Frame: Throughout the study period, 12 months ± 14 days
Population: Additional evaluations for bleeding episodes in the intent-to-treat analysis dataset: consists of all participants with at least 1 bleeding episode treated with investigational product.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Units Other Than Participants: Bleeding episodes
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 17 | 12
Number analyzed (Bleeding episodes) | 522 | 158
Scores on a scale
  Pre-Infusion (N= 513, 130) | 29.0 (43.0) [12.0 to 55.0] | 49.5 (46.9) [34.7 to 81.6]
  6 ± 0.5 hours post-infusion (N= 522, 158) | 10.0 (33.0) [4.0 to 37.0] | 33.8 (44.6) [8.0 to 52.6]
  24 ± 1 hours post-infusion (N= 512,131) | 3.0 (13.0) [1.0 to 14.0] | 6.2 (19.0) [1.0 to 20.0]
  Change (Pre-Inf to 6h post-inf) (N= 509, 129) | 10.0 [4.0 to 21.8] | 19.4 [5.0 to 41.6]
  Change (Pre-Inf to 24h post-inf) (N= 489, 102) | 18.0 [8.0 to 39.6] | 37.8 [17.0 to 75.5]

8. Secondary Outcome: Assessment of Clinical Symptoms - Visual Analog Scale (VAS): Pain in Pediatrics (<12 Years Old)
Description: Pain caused by a bleeding episode (BE) in pediatric participants (<12 years old) was measured at pre-infusion (pre-inf) and at 6 ± 0.5 h and 24 ± 1 h post-infusion (post-inf) (after the last infusion given to treat a bleeding episode) using the children's VAS pain scale (a facial expression scale with one end marked as no pain and the opposite end marked as the worst possible pain). For analysis purposes, if short acting analgesics (duration of activity approximately 6 ± 0.5 h) were used, pain was assigned the highest possible score (worst possible pain). Scores on the children's VAS scale are presented as: -No Pain -Mild Pain -Moderate pain -Severe pain -Very severe pain
Time Frame: 12 months ± 14 days
Population: as for outcome 7
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes (BEs)
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 2 | 2
Number analyzed (Bleeding episodes (BEs)) | 77 | 9
Bleeding episodes
  Pre-Infusion (N= 54, 8) - No Pain | 27 | 3
  Pre-Infusion (N= 54, 8) - Mild Pain | 3 | 1
  Pre-Infusion (N= 54, 8) - Moderate Pain | 12 | 3
  Pre-Infusion (N= 54, 8) - Severe Pain | 10 | 1
  Pre-Infusion (N= 54, 8) - Very Severe Pain | 2 | 0
  6 ± 0.5 h post-infusion (N= 74, 8) - No Pain | 47 | 3
  ± 0.5 h post-infusion (N= 74, 8) - Mild Pain | 9 | 3
  ± 0.5 h post-infusion (N= 74, 8) - Moderate Pain | 15 | 2
  ± 0.5 h post-infusion (N= 74, 8) - Severe Pain | 3 | 0
  ± 0.5 h post-infusion (N= 74, 8)- Very Severe Pain | 0 | 0
  24 ± 1 h post-infusion (N= 77, 9) - No Pain | 60 | 7
  24 ± 1 h post-infusion (N= 77, 9) - Mild Pain | 11 | 1
  24 ± 1 h post-infusion (N= 77, 9) - Moderate Pain | 6 | 1
  24 ± 1 h post-infusion (N= 77, 9) - Severe Pain | 0 | 0
  24± 1h post-infusion (N = 77, 9) -Very Severe Pain | 0 | 0

9. Secondary Outcome: Assessment of Clinical Symptoms - Range of Motion (ROM)
Description: ROM was measured using a goniometer for 3 key joints (ie, ankles, knees, and elbows) at screening, month 6, and termination (end of study visit)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
degrees
  Left Elbow - Extension: Screening | 15.0 [0.0 to 45.0] | 10.0 [0.0 to 25.0]
  Left Elbow - Extension: Month 6 (n = 18,16) | 10.0 [0.0 to 41.0] | 8.0 [0.0 to 42.5]
  Left Elbow - Extension: Termination (n = 17,16) | 20.0 [0.0 to 41.0] | 15.5 [0.0 to 40.0]
  Left Elbow - Flexion: Screening (n = 19,17) | 125.0 [90.0 to 140.0] | 115.0 [80.0 to 140.0]
  Left Elbow - Flexion: Month 6 (n = 18,16) | 130.0 [90.0 to 140.0] | 125.0 [72.5 to 143.0]
  Left Elbow - Flexion: Termination (n = 17,16) | 110.0 [90.0 to 140.0] | 125.0 [75.0 to 145.0]
  Left Elbow - Pronation: Screening (n = 18,16) | 64.0 [55.0 to 90.0] | 55.0 [22.5 to 77.5]
  Left Elbow - Pronation: Month 6 (n = 17,14) | 80.0 [60.0 to 90.0] | 67.5 [35.0 to 80.0]
  Left Elbow - Pronation: Termination (n = 17,15) | 68.0 [60.0 to 90.0] | 65.0 [30.0 to 80.0]
  Left Elbow - Supination: Screening (n = 18,16) | 75.0 [50.0 to 90.0] | 42.5 [17.5 to 77.5]
  Left Elbow - Supination: Month 6 (n = 17,14) | 80.0 [50.0 to 90.0] | 60.0 [35.0 to 80.0]
  Left Elbow - Supination: Termination (n = 17,15) | 70.0 [50.0 to 90.0] | 70.0 [35.0 to 80.0]
  Right Elbow - Extension: Screening (n = 19,17) | 20.0 [0.0 to 50.0] | 10.0 [0.0 to 50.0]
  Right Elbow - Extension: Month 6 (n = 18,16) | 17.5 [0.0 to 50.0] | 10.0 [0.0 to 42.5]
  Right Elbow - Extension: Termination (n = 18,16) | 22.5 [0.0 to 45.0] | 20.0 [0.0 to 62.5]
  Right Elbow - Flexion: Screening (n = 19,17) | 120.0 [105.0 to 140.0] | 100.0 [80.0 to 130.0]
  Right Elbow - Flexion: Month 6 (n = 18,16) | 122.5 [110.0 to 140.0] | 100.0 [85.0 to 136.0]
  Right Elbow - Flexion: Termination (n = 18,16) | 121.0 [110.0 to 140.0] | 99.0 [70.0 to 127.5]
  Right Elbow - Pronation: Screening (n = 18,16) | 75.0 [55.0 to 90.0] | 57.5 [27.5 to 80.0]
  Right Elbow - Pronation: Month 6 (n = 17,14) | 80.0 [55.0 to 90.0] | 72.5 [40.0 to 80.0]
  Right Elbow - Pronation: Termination (n = 18,15) | 67.5 [55.0 to 90.0] | 70.0 [40.0 to 80.0]
  Right Elbow - Supination: Screening (n = 18,16) | 75.0 [45.0 to 90.0] | 52.5 [20.0 to 80.0]
  Right Elbow - Supination: Month 6 (n = 17,14) | 70.0 [45.0 to 90.0] | 72.5 [30.0 to 80.0]
  Right Elbow - Supination: Termination (n = 18,15) | 75.0 [45.0 to 90.0] | 70.0 [30.0 to 80.0]
  Left Knee - Extension: Screening (n = 18,16) | 15.0 [5.0 to 90.0] | 1.5 [0.0 to 55.5]
  Left Knee - Extension: Month 6 (n = 17,14) | 15.0 [5.0 to 70.0] | 0.0 [0.0 to 20.0]
  Left Knee - Extension: Termination (n = 18,15) | 15.0 [5.0 to 90.0] | 0.0 [0.0 to 70.0]
  Left Knee - Flexion: Screening (n = 19,17) | 100.0 [80.0 to 130.0] | 90.0 [65.0 to 115.0]
  Left Knee - Flexion: Month 6 (n = 18,16) | 112.5 [80.0 to 130.0] | 97.5 [65.0 to 125.0]
  Left Knee - Flexion: Termination (n = 18,16) | 105.0 [60.0 to 130.0] | 92.5 [70.0 to 125.0]
  Right Knee - Extension: Screening (n = 18,16) | 35.0 [10.0 to 90.0] | 5.0 [0.0 to 30.0]
  Right Knee - Extension: Month 6 (n = 17,14) | 20.0 [10.0 to 90.0] | 10.0 [2.0 to 30.0]
  Right Knee - Extension: Termination (n = 18,15) | 17.5 [10.0 to 90.0] | 5.0 [0.0 to 30.0]
  Right Knee - Flexion: Screening (n = 19,17) | 90.0 [20.0 to 122.0] | 80.0 [60.0 to 125.0]
  Right Knee - Flexion: Month 6 (n = 18,16) | 90.0 [20.0 to 130.0] | 82.5 [56.0 to 127.5]
  Right Knee - Flexion: Termination (n = 18,16) | 85.0 [20.0 to 120.0] | 87.5 [56.0 to 127.5]
  Left Ankle - Dorsiflexion: Screening (n = 18,16) | 20.0 [15.0 to 30.0] | 17.5 [9.0 to 37.5]
  Left Ankle - Dorsiflexion: Month 6 (n = 17,14) | 20.0 [11.0 to 35.0] | 17.5 [8.0 to 50.0]
  Left Ankle - Dorsiflexion: Termination (n = 17,15) | 15.0 [11.0 to 25.0] | 20.0 [5.0 to 50.0]
  Left Ankle - Plantarflexion: Screening (n = 18,16) | 34.5 [30.0 to 40.0] | 30.0 [10.0 to 35.0]
  Left Ankle - Plantarflexion: Month 6 (n = 17,14) | 34.0 [25.0 to 35.0] | 30.0 [15.0 to 40.0]
  Left Ankle - Plantarflexion: Termination (n=17,15) | 35.0 [30.0 to 40.0] | 30.0 [15.0 to 35.0]
  Left Ankle - Pronation: Screening (n = 19,17) | 14.0 [10.0 to 20.0] | 15.0 [10.0 to 15.0]
  Left Ankle - Pronation: Month 6 (n = 18,15) | 15.0 [10.0 to 20.0] | 15.0 [10.0 to 16.0]
  Left Ankle - Pronation: Termination (n = 18,16) | 15.0 [10.0 to 20.0] | 12.5 [10.0 to 15.5]
  Left Ankle - Supination: Screening (n = 19,17) | 25.0 [10.0 to 30.0] | 15.0 [10.0 to 27.0]
  Left Ankle - Supination: Month 6 (n = 18,15) | 25.0 [20.0 to 30.0] | 25.0 [10.0 to 30.0]
  Left Ankle - Supination: Termination (n = 18,16) | 25.0 [16.0 to 30.0] | 20.0 [10.0 to 27.5]
  Right Ankle - Dorsiflexion: Screening (n = 18,16) | 15.0 [10.0 to 20.0] | 20.0 [7.5 to 35.0]
  Right Ankle - Dorsiflexion: Month 6 (n = 17,14) | 15.0 [15.0 to 20.0] | 25.0 [6.0 to 40.0]
  Right Ankle - Dorsiflexion: Termination (n= 17,15) | 15.0 [14.0 to 20.0] | 20.0 [10.0 to 40.0]
  Right Ankle - Plantarflexion: Screening (n= 18,16) | 35.0 [30.0 to 40.0] | 20.0 [9.0 to 39.0]
  Right Ankle - Plantarflexion: Month 6 (n= 17,14) | 30.0 [25.0 to 40.0] | 23.0 [10.0 to 40.0]
  Right Ankle - Plantarflexion: Termination(n=17,15) | 30.0 [25.0 to 40.0] | 21.0 [10.0 to 40.0]
  Right Ankle - Pronation: Screening (n = 19,17) | 10.0 [10.0 to 15.0] | 10.0 [10.0 to 20.0]
  Right Ankle - Pronation: Month 6 (n= 18,15) | 10.0 [10.0 to 20.0] | 10.0 [10.0 to 20.0]
  Right Ankle - Pronation: Termination (n= 18,16) | 10.0 [10.0 to 17.0] | 11.0 [10.0 to 17.5]
  Right Ankle - Supination: Screening (n = 19,17) | 17.0 [10.0 to 30.0] | 20.0 [10.0 to 30.0]
  Right Ankle - Supination: Month 6 (n= 18,15) | 20.0 [10.0 to 30.0] | 20.0 [10.0 to 30.0]
  Right Ankle - Supination: Termination (n= 18,16) | 20.0 [10.0 to 30.0] | 20.0 [10.0 to 30.0]

10. Secondary Outcome: Assessment of Hemostasis for Treatment of Bleeding Episodes- Overall Efficacy Rating at 6 Hours
Description: Number of rAHF-PFM-treated bleeding episodes with an assessment of hemostasis (4-point ordinal scale): Excellent: Full pain relief & bleeding cessation within ~6 hours of 1 infusion. Additional infusions may have been given to maintain hemostasis; Good: Definite pain relief and/or improvement in bleeding within ~6 hours after infusion. Possibly requires >1 infusion for complete resolution; Fair: Probable or slight relief of pain & slight improvement in bleeding within ~6 hours after infusion. Requires >1 infusion for complete resolution; None: No improvement or condition worsens
Time Frame: 6 h ± 30 min post-infusion
Population: Bleeding Episodes Analysis Set Consists of all participants who experienced a bleeding episode (BE)
Measure: Number; unit: bleeding episodes
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 14
bleeding episodes
  Excellent (n = 16, 5) | 109 | 16
  Good (n = 19, 14) | 355 | 106
  Fair (n = 15, 6) | 142 | 42
  None (n = 6, 2) | 14 | 5
  Rating Not Done (n = 3, 2) | 3 | 2
  Not Available (n = 0, 1) | 0 | 2

11. Secondary Outcome: Assessment of Hemostasis for Treatment of Bleeding Episodes- Overall Efficacy Rating at 24 Hours
Description: Number of rAHF-PFM-treated bleeding episodes with an assessment of hemostasis (4-point ordinal scale): Excellent: Full pain relief & bleeding cessation within ~24 hours of 1 infusion. Additional infusions may have been given to maintain hemostasis; Good: Definite pain relief and/or improvement in bleeding within ~24 hours after infusion. Possibly requires >1 infusion for complete resolution; Fair: Probable or slight relief of pain & slight improvement in bleeding within ~24 hours after infusion. Requires >1 infusion for complete resolution; None: No improvement or condition worsens
Time Frame: 24 ± 1 h post-infusion
Population: Bleeding Episodes Analysis Set Consists of all participants who experienced a bleeding episode (BE)
Measure: Number; unit: bleeding episodes
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 14
bleeding episodes
  Excellent (n = 16, 6) | 282 | 42
  Good (n = 19, 14) | 280 | 89
  Fair (n = 9, 3) | 36 | 12
  None (n = 1,0) | 1 | 0
  Rating Not Done (n = 8, 3) | 24 | 28
  Not Available (n = 0, 1) | 0 | 2

12. Secondary Outcome: Total Weight Adjusted Dose to Control a Bleeding Episode
Time Frame: 12 months ± 14 days
Population: Additional Evaluations for Bleeding Episodes Analysis Set - Consists of all participants with at least 1 bleeding episode treated with investigational product, FEIBA NF.
Measure: Median (Inter-Quartile Range); unit: Units/kg
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 14
Units/kg | 4049.7 [2324.5 to 7408.4] | 1524.9 [293.2 to 2883.5]
Statistical Analysis 1: Comparison: On-demand Arm vs Prophylaxis Arm; Test type: Superiority or Other; p = 0.0067, Mann-Whitney tests (Wilcoxon-Rank Sum)

13. Secondary Outcome: The Number of Bleeding Episode (BE) Which Required 1, 2, 3, or ≥4 Infusions to Control Bleeding
Time Frame: 12 months ± 14 days
Population: as for outcome 12
Measure: Number; unit: Bleeding Episodes (BEs)
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 14
Bleeding Episodes (BEs)
  1 infusion | 352 | 98
  2 infusions | 134 | 41
  3 infusions | 62 | 13
  ≥4 infusions | 75 | 21

14. Secondary Outcome: Abnormal Activated Partial Thromboplastin Time (aPTT) Assay Results
Description: The normal reference range of values for aPTT is 22.8 - 31 seconds.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 16
seconds
  Screening visit (n= 19, 16) | 67.3 [63.1 to 75.1] | 68.5 [61.0 to 73.1]
  Month 3 (n= 14, 15) | 68.0 [62.7 to 76.2] | 62.7 [57.5 to 67.2]
  Month 6 (n= 17, 15) | 68.2 [64.6 to 72.1] | 65.6 [62.6 to 69.5]
  Month 9 (n= 17, 15) | 70.0 [64.6 to 77.9] | 68.1 [58.1 to 73.9]
  Termination visit (n= 18, 16) | 69.8 [63.4 to 75.6] | 69.4 [60.5 to 77.1]

15. Secondary Outcome: Abnormal D-Dimer Assay Results
Description: The normal reference range of values for D-dimers is <500 ng/mL.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 9 | 9
ng/mL
  Screening visit (n= 7, 6) | 862.0 [647.0 to 1035.0] | 833.5 [644.0 to 1164.0]
  Month 3 (n= 7, 8) | 690.0 [561.0 to 830.0] | 1021.5 [730.0 to 1633.5]
  Month 6 (n= 9, 8) | 969.0 [753.0 to 1103.0] | 1032.0 [652.0 to 1442.5]
  Month 9 (n= 6, 8) | 731.5 [592.0 to 1398.0] | 1121.0 [942.5 to 1448.5]
  Termination visit (n= 5, 9) | 813.0 [695.0 to 1386.0] | 1031.0 [872.0 to 1258.0]

16. Secondary Outcome: Abnormal Fibrinogen Assay Results
Description: The normal reference range of values for fibrinogen is 200-400 mg/dL.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 4 | 6
mg/dL
  Screening visit (n= 4, 6) | 428.0 [414.0 to 478.5] | 422.0 [411.0 to 428.0]
  Month 3 (n= 0, 2) | NA [NA to NA] — There were no abnormal fibrinogen assay results for this arm/group at this time point | 402.0 [199.0 to 605.0]
  Month 6 (n= 3, 1) | 415.0 [412.0 to 418.0] | 759.0 [759.0 to 759.0]
  Month 9 (n= 1, 4) | 508.0 [508.0 to 508.0] | 326.5 [183.5 to 635.5]
  Termination visit (n= 2, 2) | 456.5 [425.0 to 488.0] | 522.5 [414.0 to 631.0]

17. Secondary Outcome: Abnormal Fibrin Degradation Products (FDP) Assay Results
Description: The normal reference range of values for FDP is 0-5 ug/mL.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 3 | 2
ug/mL
  Screening visit (n= 1, 2) | 16.0 [16.0 to 16.0] | 12.0 [8.0 to 16.0]
  Month 3 (n= 0, 2) | NA [NA to NA] — There were no abnormal fibrin degradation products assay results for this arm/group at this time point | 8.0 [8.0 to 8.0]
  Month 6 (n= 1, 1) | 8.0 [8.0 to 8.0] | 8.0 [8.0 to 8.0]
  Month 9 (n= 1, 2) | 8.0 [8.0 to 8.0] | 8.0 [8.0 to 8.0]
  Termination visit (n= 3, 1) | 8.0 [8.0 to 8.0] | 8.0 [8.0 to 8.0]

18. Secondary Outcome: Abnormal Prothrombin Fragment F 1.2 Assay Results
Description: The normal reference range of values for prothrombin fragment F 1.2 is 69-229 pmol/L.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 6 | 9
pmol/L
  Screening visit (n= 2, 1) | 284.0 [278.0 to 290.0] | 308.0 [308.0 to 308.0]
  Month 3 (n= 6, 7) | 336.5 [267.0 to 414.0] | 579.0 [354.0 to 972.0]
  Month 6 (n= 3, 9) | 448.0 [272.0 to 714.0] | 430.0 [366.0 to 504.0]
  Month 9 (n= 4, 9) | 382.0 [313.0 to 405.5] | 415.0 [272.0 to 472.0]
  Termination visit (n= 4, 7) | 252.5 [250.0 to 265.0] | 643.0 [376.0 to 1679.0]

19. Secondary Outcome: Abnormal Prothrombin Time Assay Results
Description: The normal reference range of values for PT is 9.7-12.3 sec.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 1 | 1
seconds
  Screening visit (n= 1, 1) | 9.4 [9.4 to 9.4] | 9.6 [9.6 to 9.6]
  Month 3 (n= 1, 0) | 9.5 [9.5 to 9.5] | NA [NA to NA] — There were no abnormal prothrombin time assay results for this arm/group at this time point
  Month 6 (n= 0, 1) | NA [NA to NA] — There were no abnormal prothrombin time assay results for this arm/group at this time point | 12.5 [12.5 to 12.5]
  Month 9 (n= 1, 1) | 12.7 [12.7 to 12.7] | 13.6 [13.6 to 13.6]
  Termination visit (n= 0, 1) | NA [NA to NA] — There were no abnormal prothrombin time assay results for this arm/group at this time point | 13.4 [13.4 to 13.4]

20. Secondary Outcome: Abnormal Thrombin-Antithrombin III (TAT) Assay Results
Description: The normal reference range of values for TAT is 1-4.1 ug/L.
Time Frame: Screening visit, Month 3, Month 6, Month 9, and Termination visit
Population: Safety Analysis Set Participants with Clinically Significant Laboratory Results
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 4 | 7
ug/L
  Screening visit (n= 4, 1) | 5.1 [4.4 to 5.9] | 5.6 [5.6 to 5.6]
  Month 3 (n= 3, 7) | 4.7 [4.5 to 5.9] | 12.3 [4.4 to 40.8]
  Month 6 (n= 3, 6) | 7.9 [6.3 to 10.5] | 5.6 [4.4 to 6.1]
  Month 9 (n= 0, 3) | NA [NA to NA] — There were no abnormal Thrombin-Antithrombin III assay results for this arm/group at this time point | 6.0 [5.6 to 52.9]
  Termination visit (n= 2, 5) | 10.3 [8.0 to 12.5] | 5.6 [5.1 to 7.3]

21. Secondary Outcome: Viral Serology From Screening Visit and Study Termination Visit: Hepatitis A, Hepatitis B, and Hepatitis C
Description: -Hepatitis A Virus Antibody (HAV Ab) -Hepatitis B Virus Core Antibody (HBcAb) -Hepatitis B Virus Surface Antibody (HBsAb) -Hepatitis B Virus Surface Antigen (HBsAg) -Hepatitis C Virus (HCV)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
participants
  HAV Ab: Screening Negative; Termination Positive | 1 | 0
  HAV Ab: Screening Negative; Termination Negative | 8 | 11
  HAV Ab: Screening Positive; Termination Positive | 8 | 4
  HAV Ab: Screening Positive; Termination Negative | 1 | 1
  HAV Ab: Serology not available | 1 | 1
  HBcAb: Screening Negative; Termination Positive | 0 | 1
  HBcAb: Screening Negative; Termination Negative | 8 | 11
  HBcAb: Screening Positive; Termination Positive | 9 | 4
  HBcAb: Screening Positive; Termination Negative | 1 | 0
  HBcAb: Serology not available | 1 | 1
  HBsAb: Screening Negative; Termination Positive | 2 | 5
  HBsAb: Screening Negative; Termination Negative | 2 | 2
  HBsAb: Screening Positive; Termination Positive | 13 | 9
  HBsAb: Screening Positive; Termination Negative | 1 | 0
  HBsAb: Serology not available | 1 | 1
  HBsAg: Screening Negative; Termination Positive | 0 | 0
  HBsAg: Screening Negative; Termination Negative | 18 | 16
  HBsAg: Serology not available | 1 | 1
  HCV: Screening Negative; Termination Positive | 0 | 0
  HCV: Screening Negative; Termination Negative | 6 | 10
  HCV: Screening Positive; Termination Positive | 12 | 6
  HCV: Screening Positive; Termination Negative | 0 | 0
  HCV: Serology not available | 1 | 1

22. Secondary Outcome: Viral Serology From Screening Visit and Study Termination Visit: HIV-1/2 Antibody (Ab)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- On-demand: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated): FEIBA NF dose and dosing interval as prescribed by the treating physician
- Prophylaxis: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : 85 ± 15 U/kg of FEIBA NF every other day during the 12-month prophylactic period
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 19 | 17
participants
  HIV 1/2 Ab: Screen Negative; Termination Positive | 0 | 0
  HIV 1/2 Ab: Screen Negative; Termination Negative | 18 | 16
  HIV 1/2 Ab: : Serology not available | 1 | 1

23. Secondary Outcome: Viral Serology From Screening Visit and Study Termination Visit: Parvovirus B19 IgG Antibody [IV]
Description: Normal range (0 - 0.89 IV); High (> 0.89 IV) - Parvovirus B19 IgG Antibody [IV] (Parvo IgG Ab)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- On-demand: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : FEIBA NF dose and dosing interval as prescribed by the treating physician
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 19 | 17
participants
  Parvo IgG Ab: Screening High ; Termination Normal | 3 | 1
  Parvo IgG Ab: Screening High ; Termination High | 14 | 13
  Parvo IgG Ab: Screening Normal; Termination Normal | 0 | 2
  Parvo IgG Ab: Screening Normal ; Termination High | 1 | 0
  Parvo IgG Ab: Serology not available | 1 | 1

24. Secondary Outcome: Viral Serology From Screening Visit and Study Termination Visit: Parvovirus B19 IgM Antibody [IV]
Description: Normal range (0 - 0.89 IV); High (> 0.89 IV) - Parvovirus B19 IgM Antibody [IV] (Parvo IgM Ab)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 19 | 17
participants
  Parvo IgM Ab: Screening High ; Termination Normal | 0 | 0
  Parvo IgM Ab: Screening High ; Termination High | 1 | 0
  Parvo IgM Ab: Screening Normal; Termination Normal | 17 | 16
  Parvo IgM Ab: Screening Normal ; Termination High | 0 | 0
  Parvo IgM Ab: Serology not available | 1 | 1

25. Secondary Outcome: Rate of Related Adverse Events (AEs) Per Year
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Related AEs per year
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
Related AEs per year | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.979]

26. Secondary Outcome: Rate of Related Adverse Events (AEs) During or Within 1 Hour of Infusion Per Year
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Related AEs within/during 1hr per year
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
Related AEs within/during 1hr per year | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

27. Secondary Outcome: Number of Related Thromboembolic Adverse Events (AEs)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set
Measure: Number; unit: Related thromboembolic AEs
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 19 | 17
Related thromboembolic AEs | 0 | 0

28. Secondary Outcome: Absolute Changes in Inhibitor Titer of Hemophilia A Participants With Shifts in Factor VIII (FVIII) Inhibitor Titer Levels
Description: Absolute Changes in Inhibitor Titer (or no change in low or high titer status): -Inhibitor Titer went from Low (≤5 BU) to Low (≤5 BU) -Inhibitor Titer went from Low (≤5 BU) to High (>5 BU) -Inhibitor Titer went from High (>5 BU) to Low (≤5 BU) -Inhibitor Titer went from High (>5 BU) to High (>5 BU)
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set - Hemophilia A study participants
Measure: Median (Inter-Quartile Range); unit: Bethesda Units (BU)
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 17 | 16
Bethesda Units (BU)
  Screening to 3 Month- Low to High (N=2, 3) | 12.1 [12.1 to 12.1] | 4.0 [0.7 to 16.8]
  Screening to 3 Month- High to Low (N=1, 0) | 2.0 [2 to 2] | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 6 Month- Low to High (N=2, 1) | 12.9 [4.9 to 20.8] | 5.3 [5.3 to 5.3]
  Screening to 6 Month- High to Low (N=1, 0) | 3.4 [3.4 to 3.4] | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 9 Month- Low to High (N=2, 1) | 5.0 [4.3 to 5.6] | 3.7 [3.7 to 3.7]
  Screening to 9 Month- High to Low (N=0, 2) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | 2.1 [0.9 to 3.2]
  Screening to Termination- Low to High (N=2, 1) | 39.2 [3.8 to 74.7] | 5.8 [5.8 to 5.8]
  Screening to Termination- High to Low (N=1, 2) | 14.6 [14.6 to 14.6] | 3.3 [3.3 to 3.3]

29. Secondary Outcome: Absolute Changes in Inhibitor Titer of Hemophilia B Participants With Shifts in Factor IX (FIX) Inhibitor Titer Levels
Description: as for outcome 28
Time Frame: 12 months ± 14 days
Population: Safety Analysis Set - Hemophilia B study participants
Measure: Median (Inter-Quartile Range); unit: Bethesda Units (BU)
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 1 | 1
Bethesda Units (BU)
  Screening to 3 Month- Low to Low (N=1, 0) | 3.2 [3.2 to 3.2] | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 3 Month- Low to High (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 3 Month- High to Low (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 3 Month- High to High (N=1, 1) | 0.3 [0.3 to 0.3] | 10.7 [10.7 to 10.7]
  Screening to 6 Month- Low to Low (N=1, 0) | 1.5 [1.5 to 1.5] | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 6 Month- Low to High (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 6 Month- High to Low (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 6 Month- High to High (N=1, 1) | 1.7 [1.7 to 1.7] | 23.2 [23.2 to 23.2]
  Screening to 9 Month- Low to Low (N=1, 0) | 3.2 [3.2 to 3.2] | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 9 Month- Low to High (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 9 Month- High to Low (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to 9 Month- High to High (N=0, 1) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | 37.0 [37.0 to 37.0]
  Screening to Termination - Low to Low (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to Termination- Low to High (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to Termination- High to Low (N=0, 0) | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point | NA [NA to NA] — There were no inhibitor titer shifts for this arm/group at this time point
  Screening to Termination - High to High (N=1, 1) | 11.3 [11.3 to 11.3] | 21.4 [21.4 to 21.4]

30. Secondary Outcome: Pharmacoeconomics: Annual Days Lost Due to Bleeding (Work or School)
Time Frame: 12 months ± 14 days
Population: Intent to Treat Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 17 | 16
days | 16.4 (25.76) [0.0 to 20.0] | 8.8 (14.42) [0.0 to 10.5]

31. Secondary Outcome: Pharmacoeconomics: Annual Number of Hospitalizations for Bleeding
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
hospitalizations | 0.6 (1.15) [0.0 to 1.0] | 0.6 (2.03) [0.0 to 0.0]

32. Secondary Outcome: Pharmacoeconomics: Annual Number of Hospitalizations for Indwelling Line
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
hospitalizations | 0.1 (0.32) [0.0 to 0.0] | 0.1 (0.25) [0.0 to 0.0]

33. Secondary Outcome: Pharmacoeconomics: Annual Number of Emergency Room Visits
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: Emergency room visits
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
Emergency room visits | 0.4 (0.98) [0.0 to 0.0] | 0.4 (1.09) [0.0 to 0.0]

34. Secondary Outcome: Pharmacoeconomics: Annual Number of Physician's Office Visits
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: Physician's office visits
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
Physician's office visits | 2.2 (4.15) [0.0 to 3.0] | 2.6 (4.60) [0.0 to 4.0]

35. Secondary Outcome: Pharmacoeconomics: Annual Total Length of Hospitalization for Bleeding
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
Days | 5.0 (9.48) [0.0 to 9.0] | 5.3 (17.00) [0.0 to 0.0]

36. Secondary Outcome: Pharmacoeconomics: Annual Total Length of Hospitalization for Indwelling Line
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 18 | 16
Days | 0.7 (2.61) | 0.7 (2.75)

37. Secondary Outcome: Pharmacoeconomics: Annual Total Number of Days Lost (Work or School)
Time Frame: 12 months ± 14 days
Population: Pharmacoeconomic Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 17 | 16
Days | 17.4 (25.42) | 15.4 (24.28)

38. Secondary Outcome: Health-Related Quality of Life (HRQoL): EuroQoL (Quality of Life)-5 Dimensions (EQ-5D) Index Scores
Description: EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome. EQ-5D Index scores based on EQ-5D questionnaire were calculated for participants ≥14 years of age, at screening, 6 months, and at termination visit. Changes in scores at 6 months and termination were also calculated. A relatively higher score represents better quality of life.
Time Frame: 12 months ± 14 days
Population: HRQoL Intent-to-Treat Analysis Dataset - comprised of all participants ≥14 years of age who were randomized, had any available assessments at any available study visits (baseline, 6- month, and 12-month) as defined in the protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 16 | 12
Scores on a scale
  Screening (N= 16, 12) | 0.627 (0.2067) | 0.620 (0.1841)
  6 Months (N= 15, 11) | 0.621 (0.1880) | 0.729 (0.1392)
  Termination (N= 15, 10) | 0.605 (0.2146) | 0.700 (0.1233)
  Change (Screening - Month 6) (N= 15, 11) | -0.006 (0.2088) | -0.096 (0.2403)
  Change (Screening - Termination) (N= 15, 10) | 0.010 (0.2470) | -0.075 (0.2594)
  Change (Month 6 - Termination) (N= 15, 10) | 0.016 (0.1765) | 0.001 (0.1493)

39. Secondary Outcome: Hemophilia-specific Quality of Life Questionnaire for Adults (Haem-A-QoL) ≥ 16 Years Old
Description: The Haem-A-QoL instrument has been developed and used in Hemophilia A patients. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. The areas covered by this instrument are: Physical Health (PH), Sports & Leisure (S&L), School & Work (W&S), Dealing with Hemophilia (Dealing), Family Planning (FP), Feeling, Relationships (R'ships), Treatment, View, and Outlook for the Future (Future). A Haem-A-QoL Total Score (Total) was also calculated. For the Haem-A-QoL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100. Haem-A-QoL scores at screening, 6 months, and at termination visit were collected. Changes in scores at 6 months and termination were also calculated.
Time Frame: 12 months ± 14 days
Population: Health-Related Quality of Life (HRQoL) Intent-to-Treat Analysis Dataset for all participants ≥ 16 years old who were randomized, had any available assessments at any available study visits (baseline, 6-month, and 12-month) as defined in the protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 15 | 12
Scores on a scale
  Dealing- Screening (N=15, 12) | 35.0 (19.72) | 26.0 (15.84)
  Dealing- Month 6 (N=14, 11) | 25.0 (16.67) | 18.9 (21.11)
  Dealing- Termination (N=14, 11) | 25.6 (25.21) | 23.7 (22.15)
  Dealing- Change (Screening - Month 6) (N=14, 11) | 10.7 (18.61) | 3.4 (22.62)
  Dealing- Change(Screening - Termination)(N=14, 11) | 10.1 (27.19) | -1.4 (21.37)
  Dealing- Change (Month 6 - Termination)(N=14, 11) | -0.6 (16.81) | -4.8 (21.26)
  FP- Screening (N=9, 8) | 16.7 (20.49) | 34.9 (31.31)
  FP- Month 6 (N=12, 7) | 20.5 (26.71) | 14.3 (11.25)
  FP- Termination (N=13, 8) | 19.1 (16.25) | 21.1 (22.14)
  FP- Change (Screening - Month 6) (N=9, 7) | -3.7 (26.94) | 14.9 (28.73)
  FP- Change(Screening - Termination)(N=9, 7) | -2.5 (25.57) | 13.1 (20.26)
  FP- Change (Month 6 - Termination)(N=11, 6) | -0.8 (32.68) | -8.3 (28.41)
  Feeling- Screening (N=15, 12) | 39.6 (28.22) | 48.2 (29.02)
  Feeling- Month 6 (N=14, 11) | 33.9 (28.77) | 29.0 (17.29)
  Feeling- Termination (N=14, 11) | 30.8 (28.53) | 26.1 (20.69)
  Feeling- Change (Screening - Month 6) (N=14, 11) | 4.9 (27.75) | 17.3 (34.72)
  Feeling- Change(Screening - Termination)(N=14, 11) | 8.0 (31.91) | 20.2 (24.58)
  Feeling- Change (Month 6 - Termination)(N=14, 11) | 3.1 (16.40) | 2.8 (23.94)
  Future- Screening (N=14, 12) | 46.8 (28.46) | 48.6 (23.32)
  Future- Month 6 (N=14, 11) | 40.2 (26.14) | 46.0 (18.03)
  Future- Termination (N=14, 11) | 47.9 (25.47) | 46.8 (18.74)
  Future- Change (Screening - Month 6) (N=13, 11) | 4.0 (26.84) | 1.1 (24.34)
  Future- Change(Screening - Termination)(N=13, 11) | -3.8 (20.53) | 0.3 (16.58)
  Future- Change (Month 6 - Termination)(N=14, 11) | -7.7 (20.25) | -0.8 (16.30)
  PH- Screening (N=15, 12) | 64.0 (22.46) | 66.4 (24.21)
  PH- Month 6 (N=14, 11) | 50.8 (27.55) | 43.1 (25.24)
  PH- Termination (N=14, 11) | 56.1 (24.98) | 42.3 (18.86)
  PH- Change (Screening - Month 6) (N=14, 11) | 14.6 (21.70) | 21.1 (28.77)
  PH- Change(Screening - Termination)(N=14, 11) | 9.3 (23.93) | 21.9 (24.79)
  PH- Change (Month 6 - Termination)(N=14, 11) | -5.3 (10.65) | 0.8 (20.20)
  R'ships- Screening (N=15, 11) | 28.3 (36.57) | 26.9 (28.83)
  R'ships- Month 6 (N=14, 11) | 19.0 (28.20) | 15.2 (13.85)
  R'ships- Termination (N=14, 10) | 17.9 (22.13) | 15.0 (17.48)
  R'ships- Change (Screening - Month 6) (N=14, 10) | 7.7 (34.04) | 10.4 (27.45)
  R'ships- Change(Screening - Termination)(N=14, 10) | 8.9 (30.57) | 12.1 (25.49)
  R'ships- Change (Month 6 - Termination)(N=14, 10) | 1.2 (21.40) | 1.7 (16.57)
  S&L- Screening (N=12, 8) | 69.3 (17.11) | 83.1 (14.13)
  S&L- Month 6 (N=12, 8) | 63.1 (23.09) | 69.7 (19.75)
  S&L- Termination (N=12, 8) | 72.3 (17.30) | 78.1 (12.52)
  S&L- Change (Screening - Month 6) (N=9, 5) | 9.9 (19.75) | 20.5 (27.97)
  S&L- Change(Screening - Termination)(N=9, 5) | 1.2 (15.91) | 7.0 (21.68)
  S&L- Change (Month 6 - Termination)(N=11, 7) | -10.2 (13.44) | -2.5 (15.61)
  Treatment- Screening (N=15, 12) | 36.9 (13.32) | 39.6 (20.70)
  Treatment- Month 6 (N=14, 11) | 30.4 (19.82) | 40.9 (16.96)
  Treatment- Termination (N=14, 11) | 34.8 (14.87) | 42.6 (17.80)
  Treatment- Change (Screening - Month 6) (N=14, 11) | 6.5 (23.72) | 0.0 (16.74)
  Treatment-Change(Screening -Termination)(N=14, 11) | 2.1 (17.81) | -1.7 (23.86)
  Treatment- Change (Month 6- Termination)(N=14, 11) | -4.4 (15.07) | -1.7 (18.70)
  View- Screening (N=15, 12) | 52.3 (24.49) | 55.6 (11.97)
  View- Month 6 (N=14, 11) | 44.3 (27.66) | 40.0 (13.23)
  View- Termination (N=14, 11) | 47.9 (22.59) | 37.7 (21.26)
  View- Change (Screening - Month 6) (N=14, 11) | 7.5 (23.68) | 14.3 (17.25)
  View- Change (Screening -Termination)(N=14, 11) | 3.9 (23.79) | 16.6 (15.01)
  View- Change (Month 6- Termination)(N=14, 11) | -3.6 (17.03) | 2.3 (20.78)
  W&S-Screening (N=13, 10) | 43.8 (25.90) | 57.7 (17.87)
  W&S- Month 6 (N=13, 9) | 31.7 (26.82) | 37.5 (20.73)
  W&S- Termination (N=12, 9) | 28.6 (22.53) | 36.8 (19.63)
  W&S- Change (Screening - Month 6) (N=12, 8) | 10.9 (30.98) | 25.3 (25.60)
  W&S- Change (Screening -Termination)(N=12, 8) | 16.1 (33.86) | 25.3 (19.01)
  W&S- Change (Month 6- Termination)(N=12, 9) | 5.2 (15.95) | 0.7 (21.75)
  Total- Screening (N=14, 12) | 44.0 (15.50) | 49.2 (15.43)
  Total- Month 6 (N=14, 11) | 37.4 (19.37) | 38.1 (11.34)
  Total- Termination (N=14, 11) | 40.2 (17.55) | 38.7 (14.21)
  Total- Change (Screening - Month 6) (N=13, 11) | 9.2 (18.44) | 10.2 (17.84)
  Total- Change (Screening -Termination)(N=13, 11) | 6.1 (15.41) | 9.5 (12.77)
  Total- Change (Month 6- Termination)(N=14, 11) | -2.7 (9.21) | -0.7 (14.40)

40. Secondary Outcome: Hemophilia-specific Quality of Life Questionnaire for Children and Adolescents < 16 Years Old (Haemo-QoL) - Parent's Evaluation
Description: The Haemo-QoL is a quality of life (QoL) assessment instrument for children and adolescents with haemophilia. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. The areas covered by this instrument are: Physical Health (PH), Sports & School (S&S), Dealing with Hemophilia (Dealing), Family, Feeling, Relationships (R'ships), Treatment, View, Outlook for the Future (Future), Friends, Others, and Support. A Haemo-QoL Total Score (Total) was also calculated. For the Haemo-QoL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100. Haemo-QoL scores at screening, 6 months, and at termination visit were collected. Changes in scores at 6 months and termination were also calculated.
Time Frame: 12 months ± 14 days
Population: Health-Related Quality of Life (HRQoL) Intent-to-Treat Analysis Dataset - for all participants <16 years old who were randomized, had any available assessments at any available study visits (baseline, 6-month, and 12-month) as defined in the protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 4 | 5
Scores on a scale
  Dealing- Screening (N=4, 4) | 25.9 (11.80) | 39.3 (17.00)
  Dealing- Month 6 (N=4, 4) | 25.6 (19.31) | 36.6 (16.07)
  Dealing- Termination (N=4, 5) | 21.4 (16.24) | 28.6 (13.36)
  Dealing- Change (Screening - Month 6) (N=4, 4) | 0.3 (8.61) | 2.7 (7.92)
  Dealing- Change(Screening - Termination)(N=4, 4) | 4.5 (7.92) | 13.4 (5.36)
  Dealing- Change (Month 6 - Termination)(N=4, 4) | 4.2 (11.85) | 10.7 (7.72)
  Family- Screening (N=4, 5) | 55.3 (19.05) | 50.9 (8.72)
  Family- Month 6 (N=4, 5) | 50.3 (27.65) | 49.1 (10.27)
  Family- Termination (N=4, 5) | 45.8 (31.03) | 39.8 (13.77)
  Family- Change (Screening - Month 6) (N=4, 5) | 5.0 (9.26) | 1.7 (15.65)
  Family- Change(Screening - Termination)(N=4, 5) | 9.5 (15.52) | 11.1 (19.22)
  Family- Change (Month 6 - Termination)(N=4, 5) | 4.5 (12.16) | 9.3 (5.24)
  Feeling- Screening (N=4, 5) | 44.1 (14.25) | 38.2 (2.77)
  Feeling- Month 6 (N=4, 5) | 50.3 (27.02) | 37.5 (22.21)
  Feeling- Termination (N=4, 5) | 33.6 (36.07) | 27.8 (16.97)
  Feeling- Change (Screening - Month 6) (N=4, 5) | -6.3 (24.27) | 0.7 (24.02)
  Feeling- Change(Screening - Termination)(N=4, 5) | 10.5 (27.92) | 10.5 (19.45)
  Feeling- Change (Month 6 - Termination)(N=4, 5) | 16.7 (13.85) | 9.7 (20.64)
  Friends- Screening (N=4, 5) | 35.9 (20.65) | 52.1 (17.18)
  Friends- Month 6 (N=4, 5) | 26.6 (17.95) | 36.3 (29.78)
  Friends- Termination (N=4, 5) | 34.4 (14.88) | 66.3 (20.06)
  Friends- Change (Screening - Month 6) (N=4, 5) | 9.4 (27.72) | 15.8 (21.88)
  Friends- Change(Screening - Termination)(N=4, 5) | 1.6 (17.95) | -14.2 (28.31)
  Friends- Change (Month 6 - Termination)(N=4, 5) | -7.8 (22.46) | -30.0 (31.68)
  Future- Screening (N=2, 2) | 53.1 (13.26) | 43.8 (17.68)
  Future- Month 6 (N=2, 2) | 40.6 (13.26) | 37.5 (8.84)
  Future- Termination (N=2, 2) | 31.3 (0.00) | 43.8 (8.84)
  Future- Change (Screening - Month 6) (N=2, 2) | 12.5 (0.00) | 6.3 (8.84)
  Future- Change(Screening - Termination)(N=2, 2) | 21.9 (13.26) | 0.0 (8.84)
  Future- Change (Month 6 - Termination)(N=2, 2) | 9.4 (13.26) | -6.3 (0.00)
  Others- Screening (N=4, 5) | 27.1 (34.44) | 29.2 (16.67)
  Others- Month 6 (N=4, 5) | 42.7 (39.14) | 24.2 (15.70)
  Others- Termination (N=4, 5) | 28.1 (32.87) | 25.8 (13.63)
  Others- Change (Screening - Month 6) (N=4, 5) | -15.6 (16.80) | 5.0 (20.28)
  Others- Change(Screening - Termination)(N=4, 5) | -1.0 (15.36) | 3.3 (15.98)
  Others- Change (Month 6 - Termination)(N=4, 5) | 14.6 (19.98) | -1.7 (10.87)
  PH- Screening (N=4, 5) | 58.0 (11.06) | 52.1 (23.23)
  PH- Month 6 (N=4, 5) | 53.6 (13.98) | 48.0 (17.23)
  PH- Termination (N=4, 5) | 41.1 (11.85) | 40.4 (17.02)
  PH- Change (Screening - Month 6) (N=4, 5) | 4.5 (12.16) | 4.1 (32.71)
  PH- Change(Screening - Termination)(N=4, 5) | 17.0 (17.10) | 11.8 (29.60)
  PH- Change (Month 6 - Termination)(N=4, 5) | 12.5 (22.87) | 7.7 (22.25)
  R'ships- Screening (N=2, 2) | 12.5 (17.68) | 43.8 (8.84)
  R'ships- Month 6 (N=2, 2) | 25.0 (35.36) | 43.8 (8.84)
  R'ships- Termination (N=2, 2) | 0.0 (0.00) | 37.5 (17.68)
  R'ships- Change (Screening - Month 6) (N=2, 2) | -12.5 (17.68) | 0.0 (0.00)
  R'ships-Change(Screening -Termination)(N=2, 2) | 12.5 (17.68) | 6.3 (8.84)
  R'ships- Change (Month 6- Termination)(N=2, 2) | 25.0 (35.36) | 6.3 (8.84)
  S&S- Screening (N=4, 5) | 67.1 (10.68) | 59.1 (23.73)
  S&S- Month 6 (N=4, 5) | 62.5 (7.74) | 56.5 (9.07)
  S&S- Termination (N=4, 5) | 55.6 (17.16) | 57.2 (17.29)
  S&S- Change (Screening - Month 6) (N=4, 5) | 4.6 (6.89) | 2.6 (16.32)
  S&S- Change (Screening -Termination)(N=4, 5) | 11.5 (12.02) | 1.9 (10.22)
  S&S- Change (Month 6- Termination)(N=4, 5) | 6.9 (18.07) | -0.8 (8.94)
  Support-Screening (N=4, 4) | 28.1 (25.77) | 51.6 (9.38)
  Support-Month 6 (N=4, 4) | 18.8 (29.32) | 42.2 (17.95)
  Support- Termination (N=4, 5) | 32.8 (32.02) | 48.8 (20.44)
  Support- Change (Screening - Month 6) (N=4, 4) | 9.4 (24.21) | 9.4 (10.83)
  Support- Change (Screening -Termination)(N=4, 4 | -4.7 (13.86) | 3.1 (15.73)
  Support- Change (Month 6- Termination)(N=4, 4) | -14.1 (21.27) | -6.3 (8.84)
  Treatment- Screening (N=4, 5) | 29.0 (13.23) | 64.2 (22.60)
  Treatment- Month 6 (N=4, 5) | 21.9 (6.90) | 54.8 (14.53)
  Treatment- Termination (N=4, 5) | 17.1 (22.12) | 41.0 (13.34)
  Treatment- Change (Screening - Month 6) (N=4, 5) | 7.1 (10.10) | 9.4 (13.06)
  Treatment- Change(Screening -Termination)(N=4, 5) | 11.9 (17.16) | 23.2 (16.94)
  Treatment- Change (Month 6- Termination)(N=4, 5) | 4.8 (22.47) | 13.8 (11.14)
  View-Screening (N=4, 5) | 47.4 (18.25) | 36.7 (16.94)
  View-Month 6 (N=4, 5) | 46.3 (24.45) | 36.4 (22.04)
  View- Termination (N=4, 5) | 32.8 (35.68) | 30.8 (12.85)
  View- Change (Screening - Month 6) (N=4, 5) | 1.1 (6.38) | 0.3 (7.63)
  View- Change (Screening -Termination)(N=4, 5) | 14.7 (18.62) | 5.9 (10.08)
  View- Change (Month 6- Termination)(N=4, 5) | 13.5 (13.02) | 5.6 (16.70)
  Total-Screening (N=4, 5) | 43.7 (13.67) | 48.1 (8.84)
  Total-Month 6 (N=4, 5) | 42.0 (13.84) | 42.3 (11.08)
  Total- Termination (N=4, 5) | 34.5 (21.83) | 39.5 (8.52)
  Total- Change (Screening - Month 6) (N=4, 5) | 1.7 (1.19) | 5.7 (14.97)
  Total- Change (Screening -Termination)(N=4, 5) | 9.1 (8.57) | 8.6 (8.72)
  Total- Change (Month 6- Termination)(N=4, 5) | 7.4 (8.91) | 2.8 (7.06)

41. Secondary Outcome: Hemophilia-specific Quality of Life Questionnaire for Children and Adolescents < 16 Years Old (Haemo-QoL) - Child's Evaluation
Description: as for outcome 40
Time Frame: 12 months ± 14 days
Population: Health-Related Quality of Life (HRQoL) Intent-to-Treat Analysis Dataset - comprised of all participants <16 years old, had any available assessments at any available study visits (baseline, 6-month, and 12-month) as defined in the protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 4 | 5
Scores on a scale
  Dealing- Screening (N=4, 4) | 33.0 (17.10) | 44.6 (20.72)
  Dealing- Month 6 (N=4, 4) | 21.4 (2.92) | 37.5 (13.20)
  Dealing- Termination (N=4, 5) | 25.0 (9.22) | 32.9 (12.73)
  Dealing- Change (Screening - Month 6) (N=4, 4) | 11.6 (15.26) | 7.1 (8.75)
  Dealing- Change(Screening - Termination)(N=4, 4) | 8.0 (15.26) | 14.3 (12.37)
  Dealing- Change (Month 6 - Termination)(N=4, 4) | -3.6 (6.52) | 7.1 (6.52)
  Family- Screening (N=4, 5) | 50.5 (23.94) | 35.6 (22.05)
  Family- Month 6 (N=4, 5) | 43.4 (28.78) | 36.4 (23.06)
  Family- Termination (N=4, 5) | 38.3 (21.25) | 32.5 (21.09)
  Family- Change (Screening - Month 6) (N=4, 5) | 7.0 (20.31) | -0.7 (16.38)
  Family- Change(Screening - Termination)(N=4, 5) | 12.2 (25.72) | 3.1 (15.51)
  Family- Change (Month 6 - Termination)(N=4, 5) | 5.2 (13.66) | 3.9 (12.20)
  Feeling- Screening (N=4, 5) | 54.8 (31.91) | 34.9 (12.89)
  Feeling- Month 6 (N=4, 5) | 41.4 (43.03) | 22.0 (18.68)
  Feeling- Termination (N=4, 5) | 34.4 (39.48) | 19.2 (15.39)
  Feeling- Change (Screening - Month 6) (N=4, 5) | 13.4 (16.91) | 12.9 (27.77)
  Feeling- Change(Screening - Termination)(N=4, 5) | 20.4 (11.77) | 15.7 (23.20)
  Feeling- Change (Month 6 - Termination)(N=4, 5) | 7.0 (7.79) | 2.8 (15.26)
  Friends- Screening (N=4, 5) | 34.4 (25.26) | 58.8 (20.54)
  Friends- Month 6 (N=4, 5) | 28.1 (15.73) | 42.5 (29.78)
  Friends- Termination (N=4, 5) | 32.8 (12.88) | 56.3 (27.24)
  Friends- Change (Screening - Month 6) (N=4, 5) | 6.3 (25.52) | 16.3 (24.84)
  Friends- Change(Screening - Termination)(N=4, 5) | 1.6 (28.58) | 2.5 (22.79)
  Friends- Change (Month 6 - Termination)(N=4, 5) | -4.7 (17.95) | -13.8 (20.44)
  Future- Screening (N=2, 2) | 40.6 (13.26) | 43.8 (17.68)
  Future- Month 6 (N=2, 2) | 43.8 (17.68) | 43.8 (17.68)
  Future- Termination (N=2, 2) | 46.9 (22.10) | 28.1 (22.10)
  Future- Change (Screening - Month 6) (N=2, 2) | -3.1 (4.42) | 0.0 (0.00)
  Future- Change(Screening - Termination)(N=2, 2) | -6.3 (8.84) | 15.6 (4.42)
  Future- Change (Month 6 - Termination)(N=2, 2) | -3.1 (4.42) | 15.6 (4.42)
  Others- Screening (N=4, 5) | 42.7 (33.74) | 26.7 (20.11)
  Others- Month 6 (N=4, 5) | 33.3 (40.11) | 16.7 (15.02)
  Others- Termination (N=4, 5) | 18.8 (21.11) | 13.3 (12.64)
  Others- Change (Screening - Month 6) (N=4, 5) | 9.4 (8.59) | 10.0 (25.79)
  Others- Change(Screening - Termination)(N=4, 5) | 24.0 (14.18) | 13.3 (23.09)
  Others- Change (Month 6 - Termination)(N=4, 5) | 14.6 (19.39) | 3.3 (16.24)
  PH- Screening (N=4, 5) | 67.0 (24.98) | 42.1 (32.28)
  PH- Month 6 (N=4, 5) | 49.1 (14.69) | 33.9 (16.66)
  PH- Termination (N=4, 5) | 41.1 (23.05) | 25.7 (10.83)
  PH- Change (Screening - Month 6) (N=4, 5) | 17.9 (19.56) | 8.2 (34.43)
  PH- Change(Screening - Termination)(N=4, 5) | 25.9 (14.40) | 16.4 (29.73)
  PH- Change (Month 6 - Termination)(N=4, 5) | 8.0 (12.16) | 8.2 (20.66)
  R'ships- Screening (N=2, 2) | 6.3 (8.84) | 43.8 (8.84)
  R'ships- Month 6 (N=2, 2) | 18.8 (26.52) | 43.8 (8.84)
  R'ships- Termination (N=2, 2) | 6.3 (8.84) | 18.8 (26.52)
  R'ships- Change (Screening - Month 6) (N=2, 2) | -12.5 (17.68) | 0.0 (0.00)
  R'ships-Change(Screening -Termination)(N=2, 2) | 0.0 (0.00) | 25.0 (17.68)
  R'ships- Change (Month 6- Termination)(N=2, 2) | 12.5 (17.68) | 25.0 (17.68)
  S&S- Screening (N=4, 5) | 53.3 (14.74) | 51.3 (19.82)
  S&S- Month 6 (N=4, 5) | 46.8 (13.42) | 54.2 (5.53)
  S&S- Termination (N=4, 5) | 33.2 (5.64) | 49.8 (18.49)
  S&S- Change (Screening - Month 6) (N=4, 5) | 6.5 (11.42) | -2.8 (18.53)
  S&S- Change (Screening -Termination)(N=4, 5) | 20.1 (14.74) | 1.5 (18.74)
  S&S- Change (Month 6- Termination)(N=4, 5) | 13.5 (9.10) | 4.4 (15.19)
  Support-Screening (N=4, 4) | 32.8 (3.13) | 62.5 (31.04)
  Support-Month 6 (N=4, 4) | 28.1 (10.83) | 56.3 (31.87)
  Support- Termination (N=4, 5) | 17.2 (17.21) | 65.0 (15.69)
  Support- Change (Screening - Month 6) (N=4, 4) | 4.7 (12.88) | 6.3 (31.46)
  Support- Change (Screening -Termination)(N=4, 4 | 15.6 (18.75) | -3.1 (18.75)
  Support- Change (Month 6- Termination)(N=4, 4) | 10.9 (10.67) | -9.4 (25.77)
  Treatment- Screening (N=4, 5) | 27.3 (15.38) | 69.6 (25.63)
  Treatment- Month 6 (N=4, 5) | 30.6 (16.50) | 56.8 (15.89)
  Treatment- Termination (N=4, 5) | 35.9 (26.10) | 44.2 (27.10)
  Treatment- Change (Screening - Month 6) (N=4, 5) | -3.2 (4.43) | 12.9 (21.22)
  Treatment- Change(Screening -Termination)(N=4, 5) | -8.6 (13.86) | 25.4 (28.00)
  Treatment- Change (Month 6- Termination)(N=4, 5) | -5.3 (11.25) | 12.6 (15.53)
  View-Screening (N=4, 5) | 46.0 (19.33) | 31.9 (14.36)
  View-Month 6 (N=4, 5) | 39.3 (33.02) | 32.4 (19.41)
  View- Termination (N=4, 5) | 32.5 (32.75) | 32.2 (8.60)
  View- Change (Screening - Month 6) (N=4, 5) | 6.7 (14.96) | -0.5 (18.94)
  View- Change (Screening -Termination)(N=4, 5) | 13.5 (16.56) | -0.3 (10.77)
  View- Change (Month 6- Termination)(N=4, 5) | 6.8 (8.67) | 0.2 (13.48)
  Total-Screening (N=4, 5) | 44.9 (12.28) | 45.1 (9.16)
  Total-Month 6 (N=4, 5) | 37.4 (17.91) | 37.7 (9.87)
  Total- Termination (N=4, 5) | 32.2 (17.96) | 35.3 (9.06)
  Total- Change (Screening - Month 6) (N=4, 5) | 7.5 (7.21) | 7.4 (16.57)
  Total- Change (Screening -Termination)(N=4, 5) | 12.7 (8.69) | 9.8 (12.35)
  Total- Change (Month 6- Termination)(N=4, 5) | 5.2 (3.55) | 2.5 (9.46)

42. Secondary Outcome: Health-Related Quality of Life (HRQoL) - General Pain Assessment Using a Visual Analogue Scale (VAS) in Adults and Adolescents ≥12 Years Old
Description: General pain was assessed using a VAS pain scale at screening, 6 months, and at termination. Unlike the VAS pain assessment for pain of bleeding episodes (Outcome above), this general pain assessment did not take use of analgesics into account. For the pain scale, a higher number indicates worse pain. The visual analog scale ranges from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (=0) and 'Best imaginable health state' (=100). A positive change from baseline indicates improvement. Change in VAS scores at 6 months and study termination were also compared relative to Baseline/Screening scores (ie, (Baseline/Screening VAS score) - (VAS score at 6 months and study termination).
Time Frame: Baseline, 6 months and 12 months ± 14 days
Population: Health-Related Quality of Life (HRQoL) Intent-to-Treat Analysis Dataset - comprised of all participants ≥12 years old who were randomized, had any available assessments at any available study visits (baseline, 6-month, and 12-month) as defined in the protocol
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 17 | 15
Scores on a scale
  Screening (N= 17, 15) | 35.2 (30.15) | 55.5 (23.68)
  Month 6 (N= 16, 14) | 36.6 (25.81) | 32.7 (26.24)
  Termination (N= 16, 14) | 32.4 (21.97) | 29.8 (30.48)
  Change (Screening - Month 6) (N= 16, 14) | 0.8 (31.77) | 20.3 (38.91)
  Change (Screening - Termination) (N= 16, 14) | 5.0 (28.70) | 23.2 (46.61)
  Change (Month 6 - Termination) (N= 16, 14) | 4.2 (21.82) | 2.9 (19.62)

43. Secondary Outcome: Health-Related Quality of Life (HRQoL) - General Pain Assessment Using a Visual Analogue Scale (VAS) in Pediatrics <12 Years Old
Description: General pain was assessed using the children's VAS pain scale (a facial expression scale with one end marked as no pain and the opposite end marked as the worst possible pain). Assessments were done at the screening, 6 months, and termination visits. Scores on the children's VAS scale are presented as: -No Pain -Mild Pain -Moderate pain -Severe pain -Very severe pain Unlike the VAS pain assessment for pain of bleeding episodes (Outcome above), this general pain assessment did not take use of analgesics into account. Change in VAS scores at 6 months and study termination were also compared relative to Baseline/Screening scores (ie, (Baseline/Screening VAS score) - (VAS score at 6 months and study termination).
Time Frame: Baseline, 6 months and 12 months ± 14 days
Population: Health-Related Quality of Life (HRQoL) Intent-to-Treat Analysis Dataset - comprised of all participants <12 years old who were randomized, had any available assessments at any available study visits (baseline, 6-month, and 12-month) as defined in the protocol
Measure: Number; unit: participants
Arm/Group | On-demand Arm | Prophylaxis Arm
Number analyzed (Participants) | 2 | 2
participants
  Screening - No Pain | 1 | 0
  Screening - Mild Pain | 0 | 1
  Screening - Moderate Pain | 1 | 0
  Screening - Severe Pain | 0 | 1
  Screening - Very Severe Pain | 0 | 0
  Month 6 - No Pain | 0 | 0
  Month 6 - Mild Pain | 1 | 2
  Month 6 - Moderate Pain | 1 | 0
  Month 6 - Severe Pain | 0 | 0
  Month 6 - Very Severe Pain | 0 | 0
  Termination visit - No Pain | 0 | 1
  Termination visit - Mild Pain | 0 | 0
  Termination visit - Moderate Pain | 1 | 1
  Termination visit - Severe Pain | 0 | 0
  Termination visit - Very Severe Pain | 1 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period of 3 years and 7 months
Groups:
- Prophylaxis Arm: Factor VIII Inhibitor Bypassing Activity (nanofiltered, vapor heat-treated) : 85 ± 15 U/kg of FEIBA NF every other day during the 12-month ± 14 days prophylactic period
Arm/Group | On-demand Arm | Prophylaxis Arm
Serious Adverse Events (participants affected / at risk) | 7/19 | 6/17
Other Adverse Events (participants affected / at risk) | 4/19 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-demand Arm (N=19) | Prophylaxis Arm (N=17)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematoma Infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatitis B Surface Antibody Positive (Investigations) | 1 (1) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (8)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catheter Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-demand Arm (N=19) | Prophylaxis Arm (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study: PIs may require prior written approval, or be restricted from independently publishing results until the earlier of the primary multicenter publication or ≤36 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) prior to submission for publication, and shall review and if necessary amend the manuscript in ≤60 days